CLINICAL TRIAL: NCT00744523
Title: ARMOUR: Proximal Protection With The Mo.Ma Device During Carotid Stenting
Brief Title: Proximal Protection With The Mo.Ma Device During Carotid Stenting
Acronym: ARMOUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P-2850
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Results first posted 2010-05-05 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Carotid Artery Disease
Keywords: carotid artery stenting; stroke; cerebral protection; high surgical risk
MeSH Terms: conditions — Carotid Artery Diseases; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mo.ma cerebral protection device (Experimental): Mo.Ma cerebral protection device
  Interventions: Device: Mo.Ma cerebral protection device

INTERVENTIONS:
Device: Mo.Ma cerebral protection device — Proximal embolic protection based on the principle endovascular clamping consisting of a catheter with two compliant balloons. Mo.Ma is designed to achieve cerebral protection by proximal blood flow blockage at the carotid bifurcation: antegrade and retrograde flow blockage are achieved by proximal balloon occlusion of the CCA and distal balloon occlusion of the ECA. Cerebral protection is established prior to the initial wire passage through the stenosis and maintained during the entire procedure. Mo.Ma provides withdrawal of embolic particles by allowing manual syringe aspiration of any micro-emboli at the end of the procedure before restoring blood flow through the stented vessel.
  Other Names: Mo.Ma

SUMMARY:
The objective of the ARMOUR study is to evaluate the safety and effectiveness of the Mo.Ma proximal flow blockage cerebral protection device for patients at high surgical risk for carotid endarterectomy who undergo carotid artery stenting

DETAILED DESCRIPTION:
Test Device:

Mo.Ma™ Proximal Flow Blockage Cerebral Protection Device. Single size catheter device with a 9 French introducer sheath compatible shaft (outer diameter) and a 6 French compatible working channel (inner diameter), integrating two compliant balloons intended to achieve endovascular clamping of external carotid arteries (ECA) 3-6 mm in diameter and common carotid arteries (CCA) 5-13 mm in diameter.

Primary Objective:

Evaluate the safety and effectiveness of the Mo.Ma device for cerebral protection in the treatment of internal carotid artery (ICA) stenoses, which may or may not involve the bifurcation of the CCA, in subjects considered to be at high surgical risk for complications during carotid endarterectomy (CEA).

Primary Endpoint:

Major adverse cardiac and cerebrovascular events (MACCE) within 30 days of implantation. MACCE are defined as: any myocardial infarction (MI), stroke, or death through day 30 post-procedure.

ELIGIBILITY:
General inclusion criteria Subject meets one or more of the high surgical risk criteria.

* Subject is ≥ 18 years old.
* Subject is a candidate for single lesion carotid artery stenting using a femoral arterial approach.
* Subject is willing and able to comply with follow-up evaluations at the specified times.
* Subject (or legal representative) understands the nature of the procedure and provides informed consent, prior to enrollment in the study.
* If female subject, is not currently pregnant and has stated that she has no intention of becoming pregnant during the study.

Angiographic inclusion criteria (as determined ≤ 30 days prior to procedure):

* Target lesion stenosis (% stenosis = (1-N/D) X 100)1, documented by selective angiography pre-intervention, is

  * ≥ 80% stenosis for asymptomatic subjects or
  * ≥ 50% stenosis for symptomatic subjects. Symptomatic is defined as carotid stenosis associated with ipsilateral transient or visual TIA evidenced byamaurosis fugax, ipsilateral hemispheric TIAs or ipsilateral ischemic stroke within 6 months prior to enrollment.
* Target lesion is within the internal carotid artery and/or involves the bifurcation of the CCA.
* External carotid artery diameter where the Mo.Ma device will be positioned is 3-6 mm.
* Common carotid artery diameter where the Mo.Ma device will be positioned is 5-13 mm.

General exclusion criteria

* Subject has participated in, is participating in, or plans to participate in another clinical study that may affect either the pre-procedure or follow-up results.
* Subject has chronic or paroxysmal atrial fibrillation that is not treated by Coumadin.
* Subject has undergone prior stenting of the ipsilateral carotid artery.
* Subject's life expectancy is less than twelve months.
* Subject is unable to respond to external questions and stimuli and to exert a pressure with the contralateral hand.
* Subject is suffering from dementia.
* Subject has documented intolerance to BOTH heparin and Angiomax.
* Subject has an allergy or contraindication to acetylsalicylic acid (ASA).
* Subject has a documented allergy to the device materials.
* Subject has a documented allergy to radiographic contrast that cannot be pre-treated.
* Subject has a documented allergy or contraindication to BOTH clopidogrel and ticlopidine.
* Subject has had active bleeding diathesis requiring blood transfusion within one (1) month prior to index procedure.
* Subject has had an MI within 72 hours prior to carotid stenting.
* Subject has had coronary artery bypass graft (CABG) or vascular surgery within 30 days PRIOR TO index procedure (percutaneous coronary intervention is permissible provided cardiac enzymes are normal within 24 hours of index procedure), OR has planned CABG, vascular surgery, percutaneous coronary intervention (PCI), or has other invasive medical procedures planned within 30 days AFTER index procedure.(Unplanned urgent or emergent procedures may be performed at anytime as clinically indicated).
* Subject has a major residual neurological deficit (stroke scales: Barthel ≤ 60, NIH ≥ 15 or Rankin > 3) at pre-procedure neurological exam.
* Subject has had a transient ischemic attack (TIA) or amaurosis fugax within 48 hours prior to index procedure.
* Subject has had a stroke or retinal artery occlusion within one (1) month prior to index procedure.
* Subject had abnormal pre-intervention blood counts with platelets < 50,000/cubic mm or > 700,000/cubic mm or white blood cell count < 3,000/cubic mm.
* Subject has severe chronic renal failure (creatinine > 2.5 mg/dl).
* Subject is currently being treated for cerebral carcinoma or sarcoma.
* Subject has peripheral vascular disease, which precludes safe femoral artery sheath insertion.
* Subject is unable or unwilling to undergo insertion of a temporary pacemaker.

Angiographic exclusion criteria (as determined ≤ 30 days prior to procedure):

* The target carotid artery is completely occluded.
* The common carotid artery ostium has stenosis that requires treatment.
* Multiple carotid stenoses exist in the internal carotid artery (ICA) that cannot be covered by one stent.
* The presence of ipsilateral intracranial stenosis that requires treatment.
* The presence of any intracranial tumor(s), arteriovenous malformation(s) (AVMs), or aneurysm(s) requiring treatment.
* The inability to position a stiff .035" guidewire in the external carotid artery (ECA).
* Contralateral occlusion of internal carotid artery and vertebral arteries.
* Aortic arch anatomical anomalies that preclude the safe placement of the device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Ansel, MD, Principal Investigator — Midwest Cardiology Research Foundation; L. Nelson Hopkins, MD, Principal Investigator — University at Buffalo Neurosurgery
Locations (2):
- United States (2):
  - University at Buffalo Neurosurgery, Buffalo, New York
  - MidWest Cardiology Research Foundation, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was approved to enroll subjects from a maximum of 25 (combined United States [US] and European Union [EU]) medical institutions (public and academic research center hospitals). Subjects were enrolled from September 2007 to February 2009.
Groups:
- MO.MA Roll-In Cases: All subjects who were enrolled prior to the pivotal phase of the trial at each US site. All subjects who fulfilled the eligibility criteria and were screened and enrolled to undergo carotid stenting with cerebral protection with the MO.MA proximal flow blockage cerebral protection device
- MO.MA Pivotal Subjects: All subjects who fulfilled the eligibility criteria and were screened and enrolled to undergo carotid stenting with cerebral protection with the MO.MA proximal flow blockage cerebral protection device
Period: Procedure
Arm/Group | MO.MA Roll-In Cases | MO.MA Pivotal Subjects
Started | 37 | 225
Completed | 37 | 225
Not Completed | 0 | 0
Period: 30 Days After the Procedure
Arm/Group | MO.MA Roll-In Cases | MO.MA Pivotal Subjects
Started | 37 | 225
Completed | 37 | 220
Not Completed | 0 | 5
Not completed — Insufficient follow-up | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MO.MA Roll-In Cases | MO.MA Pivotal Subjects | Total
Number analyzed (Participants) | 37 | 225 | 262
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 37 | 43
  >=65 years | 31 | 188 | 219
Age, Customized [Number; unit: participants]
  < 80 years | 26 | 160 | 186
  >= 80 years | 11 | 65 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.28 (10.38) | 74.66 (8.54) | 74.61 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 75 | 87
  Male | 25 | 150 | 175
Region of Enrollment [Number; unit: participants]
  United States | 37 | 147 | 184
  Europe | 0 | 78 | 78
History of Diabetes [Number; unit: participants]
  Yes | 15 | 83 | 98
  No | 21 | 141 | 162
  No Response | 1 | 1 | 2
History of Hypertension [Number; unit: participants]
  Yes | 32 | 196 | 228
  No | 5 | 29 | 34
Symptomatic [1] [Number; unit: participants] — [1]Presence of baseline neurological symptoms within 6 months prior to enrollment.
  participants
    Symptomatic | 8 | 34 | 42
    Asymptomatic | 29 | 191 | 220

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiac and Cerebrovascular Events (MACCE) Within 30 Days of the Procedure.
Description: Number of subjects with one or more Major Adverse Cardiac and Cerebrovascular Events through 30 days after the procedure. MACCE are defined as: any myocardial infarction (MI), stroke, or death through day 30 post-procedure.
Time Frame: Up to 30 days after the procedure was performed
Population: Roll In Population - All subjects enrolled prior to the pivotal phase at each US site. Pivotal - All subjects who fulfilled the eligibility criteria and were screened and enrolled to undergo carotid stenting with cerebral protection with the MO.MA device. ITT - All subjects enrolled regardless of subsequent treatment.
Measure: Number; unit: participants
Groups:
- MO.MA Training Cases (Roll-In): All subjects who were enrolled prior to the pivotal phase of the trial at each US site. All subjects who fulfill the eligibility criteria will be screened and enrolled to undergo carotid stenting with cerebral protection with the MO.MA proximal flow blockage cerebral protection device
- MO.MA Pivotal Subjects: All subjects who fulfilled the eligibility criteria and were screened and enrolled to undergo carotid stenting with cerebral protection with the MO.MA device.
Arm/Group | MO.MA Training Cases (Roll-In) | MO.MA Pivotal Subjects
Number analyzed (Participants) | 37 | 225
participants
  Any MACCE during 30 days after the procedure | 0 | 6
  Any myocardial infarction | 0 | 0
  Stroke | 0 | 5
  Death | 0 | 2
  Any MACCE during the procedure | 0 | 4
  Any MACCE at discharge | 0 | 4
Statistical Analysis 1: Comparison: MO.MA Training Cases (Roll-In) vs MO.MA Pivotal Subjects; The ARMOUR trial tested the null hypothesis that the MACCE rate was greater than or equal to the Performance Goal (PG) of 13% versus the alternative hypothesis that the true MACCE rate was less than the PG. The sample size was calculated based on 90% power and a Type I error rate of 0.05 (one-sided). The Performance Goal was calculated from results of carotid artery stenting trials that utilized embolic protection devices (EPD); Test type: Superiority or Other; p < 0.05, t-test, 1 sided; proportion of the primary endpoint = 2.7, 95% CI 1-sided [upper limit 5.2], Standard Error of Mean 5 — Parameter Dispersion Type of Standard Error of the mean is meant to state that 'mean" is the mean of proportions in the sense of a central-limit theorem

2. Secondary Outcome: Device Success
Description: Number of subjects in which the MO.MA was able to be positioned, deployed, and retrieved intact during the index procedure.
Time Frame: The entire duration of the index procedure
Population: Roll In Population - All subjects enrolled prior to the pivotal phase at each US site. Pivotal - All subjects who fulfilled the eligibility criteria who were screened and enrolled to undergo carotid stenting with cerebral protection with the MO.MA device. ITT - All subjects enrolled regardless of subsequent treatment.
Measure: Number; unit: participants
Arm/Group | MO.MA Roll-In Cases | MO.MA Pivotal Subjects
Number analyzed (Participants) | 37 | 225
participants | 37 | 221

3. Secondary Outcome: Technical Success
Description: Number of subjects with device success and the ability to successfully implant a carotid stent and obtain a residual stenosis < 30% during the index procedure(as evaluated by the angiographic core laboratory).
  Note: Three subjects were missing final angiographic results and therefore Technical and Procedural success could not be defined for these three subjects, thereby, decreasing the number of participants analyzed from 225 to 222.
Time Frame: The entire duration of the index procedure
Population: Roll-In participants were analysed on the number of roll-in cases performed. Pivotal subjects were analysed as Intention To Treat (ITT).
Measure: Number; unit: participants
Arm/Group | MO.MA Roll-In Cases | MO.MA Pivotal Subjects
Number analyzed (Participants) | 36 | 222
participants | 34 | 210

4. Secondary Outcome: Procedural Success
Description: Number of subjects with technical success without the occurrence of any MACCE or unresolved antegrade flow blockage intolerance during the index hospitalization.
  Note: Three subjects were missing final angiographic results and therefore Technical and Procedural success could not be defined for these three subjects, thereby, decreasing the number of participants analyzed from 225 to 222.
Time Frame: The entire duration of the index procedure through hospital discharge
Measure: Number; unit: participants
Arm/Group | MO.MA Roll-In Cases | MO.MA Pivotal Subjects
Number analyzed (Participants) | 36 | 222
participants | 33 | 207

5. Secondary Outcome: Restenosis at 30 Days
Description: Number of subjects with re-narrowing of the lesion at 30 days as defined as a >= 50% stenosis measured by duplex ultrasound scan.
Time Frame: Up to 30 days after the procedure was performed
Measure: Number; unit: participants
Arm/Group | MO.MA Roll-In Cases | MO.MA Pivotal Subjects
Number analyzed (Participants) | 34 | 190
participants | 2 | 3

6. Secondary Outcome: Target Lesion Revascularization at 30 Days
Description: Number of subjects with any repeat invasive procedure, including angioplasty, stenting, endarterectomy, or thrombolysis, performed to open or increase lumen diameter inside or within 10 mm of the previously treated lesion.
Time Frame: Up to 30 days after the procedure was performed
Measure: Number; unit: participants
Arm/Group | MO.MA Roll-In Cases | MO.MA Pivotal Subjects
Number analyzed (Participants) | 37 | 220
participants | 0 | 0

7. Secondary Outcome: Access Site Adverse Events
Description: Number of subjects with adverse events at the percutaneous access site as a result of the index procedure, including bruising, hematoma and bleeding requiring treatment by transfusion of blood products, surgical repair, ultrasound compression or thrombin injection.
Time Frame: Index Procedure through Hospital Discharge
Measure: Number; unit: participants
Arm/Group | MO.MA Roll-In Cases | MO.MA Pivotal Subjects
Number analyzed (Participants) | 37 | 225
participants | 2 | 7

ADVERSE EVENTS:
Time Frame: Index procedure through the 30 day follow-up visit.
Arm/Group | MO.MA Roll-In Cases | MO.MA Pivotal Subjects
Serious Adverse Events (participants affected / at risk) | 11/37 | 37/225
Other Adverse Events (participants affected / at risk) | 27/37 | 132/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | MO.MA Roll-In Cases (N=37) | MO.MA Pivotal Subjects (N=225)
Anaemia (Blood and lymphatic system disorders) | 0/0 (0) | 4 (4)
Blood urea increased (Investigations) | 0/0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0/0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0/0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0/0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 0/0 (0) | 1 (1)
Cerebral hyperfusion syndrome (Nervous system disorders) | 0/0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0/0 (0) | 2 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0/0 (0) | 1 (1)
Confusional state (Nervous system disorders) | 1 (1) | 0/0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0/0 (0)
Coronary artery disease (Cardiac disorders) | 0/0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0/0 (0)
Ejection fraction abnormal (Investigations) | 0/0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0/0 (0) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0/0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/0 (0) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 0/0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0/0 (0) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Hypotension (Vascular disorders) | 7 (7) | 6 (6)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0/0 (0)
Ischaemic stroke (Nervous system disorders) | 0/0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0/0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0/0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0/0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0/0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0/0 (0) | 3 (3)
Renal failure acute (Renal and urinary disorders) | 0/0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0/0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0/0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0/0 (0) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 0/0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0/0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | MO.MA Roll-In Cases (N=37) | MO.MA Pivotal Subjects (N=225)
Abdominal pain upper (Gastrointestinal disorders) | 0/0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0/0 (0)
Anaemia (Blood and lymphatic system disorders) | 0/0 (0) | 9 (9)
Angina pectoris (Cardiac disorders) | 0/0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0/0 (0)
Arterioventricular block (Cardiac disorders) | 0/0 (0) | 1 (1)
Arterioventricular block first degree (Cardiac disorders) | 0/0 (0) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0/0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 0/0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/0 (0) | 1 (1)
Bladder obstruction (Renal and urinary disorders) | 0/0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0/0 (0) | 5 (5)
Blood pressure decreased (Investigations) | 0/0 (0) | 1 (1)
Blood urea increased (Investigations) | 0/0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 6 (6) | 13 (14)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Burns first degree (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0/0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0/0 (0) | 2 (2)
Cardiac flutter (Cardiac disorders) | 0/0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0/0 (0) | 1 (1)
Carotid artery dissection (Nervous system disorders) | 0/0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery thrombosis (Nervous system disorders) | 0/0 (0) | 1 (1)
Catheter site discharge (General disorders) | 0/0 (0) | 2 (2)
Catheter site haematoma (General disorders) | 3 (3) | 2 (2)
Catheter site haemorrhage (General disorders) | 0/0 (0) | 2 (2)
Catheter site pain (General disorders) | 0/0 (0) | 1 (1)
Cerebral hyperfusion syndrome (Nervous system disorders) | 0/0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0/0 (0) | 2 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/0 (0)
Clumsiness (Nervous system disorders) | 0/0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0/0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0/0 (0) | 1 (1)
Confusional state (Nervous system disorders) | 2 (2) | 3 (3)
Convulsion (Nervous system disorders) | 1 (2) | 1 (1)
Coordination abnormal (Nervous system disorders) | 1 (1) | 0/0 (0)
Coronary artery disease (Cardiac disorders) | 0/0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0/0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0/0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0/0 (0) | 2 (2)
Disorientation (Nervous system disorders) | 0/0 (0) | 3 (3)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0/0 (0)
Dizziness (Nervous system disorders) | 0/0 (0) | 4 (4)
Dysarthia (Nervous system disorders) | 0/0 (0) | 7 (7)
Dyskinesia (Nervous system disorders) | 0/0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 5 (5)
Ear pain (Ear and labyrinth disorders) | 0/0 (0) | 1 (1)
Ejection fraction abnormal (Investigations) | 0/0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0/0 (0) | 1 (1)
Electrocardiogram ST segment abnormal (Investigations) | 0/0 (0) | 3 (3)
Electrocardiogram T wave abnormal (Investigations) | 0/0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0/0 (0) | 1 (1)
Embolism (Vascular disorders) | 0/0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 1 (1)
Epitaxis (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 1 (1)
Facial paraesis (Nervous system disorders) | 1 (1) | 0/0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0/0 (0)
Fibrosis (General disorders) | 0/0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/0 (0) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0/0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0/0 (0) | 2 (2)
Haempotysis (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 8 (9)
Hemiparesis (Nervous system disorders) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0/0 (0) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 0/0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (4) | 13 (14)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 3 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 0/0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0/0 (0) | 1 (1)
Hypotension (Vascular disorders) | 17 (18) | 51 (52)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0/0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0/0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0/0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0/0 (0) | 8 (8)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 1 (1)
Monoparesis (Nervous system disorders) | 0/0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0/0 (0) | 1 (1)
Muscular weakness (Nervous system disorders) | 1 (1) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0/0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0/0 (0)
Myocardial infarction (Cardiac disorders) | 0/0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0/0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 7 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (3)
Odynophagia (Gastrointestinal disorders) | 0/0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0/0 (0) | 1 (1)
Pain (General disorders) | 0/0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0/0 (0) | 1 (1)
Peripheral coldness (General disorders) | 0/0 (0) | 1 (1)
Pharyngeal hypoaesthesia (Nervous system disorders) | 0/0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Post operative wound infection (Infections and infestations) | 0/0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Psychotic disorder (Psychiatric disorders) | 0/0 (0) | 1 (1)
Pyrexia (General disorders) | 0/0 (0) | 2 (2)
Rales (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0/0 (0) | 3 (3)
Renal failure acute (Renal and urinary disorders) | 0/0 (0) | 3 (3)
Restlessness (Psychiatric disorders) | 0/0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0/0 (0)
Simple partial seizures (Nervous system disorders) | 0/0 (0) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 4 (4)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 8 (8)
Sinusitis (Infections and infestations) | 0/0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0/0 (0) | 5 (5)
Supraventricular extrasystoles (Cardiac disorders) | 0/0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 4 (5)
Tachycardia (Cardiac disorders) | 0/0 (0) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1) | 0/0 (0)
Tongue paralysis (Nervous system disorders) | 1 (1) | 0/0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0/0 (0) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 0/0 (0) | 2 (2)
Unresponsive to stimuli (Nervous system disorders) | 0/0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0/0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0/0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 0/0 (0) | 2 (2)
Vascular pseudoaneurysm (Vascular disorders) | 0/0 (0) | 5 (5)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0/0 (0)
Vertebral injury (Injury, poisoning and procedural complications) | 0/0 (0) | 1 (1)
Visual acuity reduced (Nervous system disorders) | 0/0 (0) | 1 (1)
Visual disturbance (Eye disorders) | 0/0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0/0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0/0 (0) | 8 (8)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days